CLINICAL TRIAL: NCT04053504
Title: Feasibility Study of Family Teamwork Peer-Delivery
Acronym: TEAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ashley Butler, Associate Professor, Pediatrics-Psychology, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-40380; DP3DK113236 (NIH)
Record Dates: First submitted 2019-07-08; First posted 2019-08-12 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Type 1 Diabetes
Keywords: Health disparities; Family teamwork; Peer-delivered intervention; Facilitators to diabetes management; Barriers to diabetes management; Community-based intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Behavioral intervention delivered by parent peer leaders.
  Interventions: Behavioral: Family Teamwork-Peer Delivery
- Standard Care (No Intervention): Standard diabetes care

INTERVENTIONS:
Behavioral: Family Teamwork-Peer Delivery — Children with T1D and their parent will participate in 6 in-person FT-P group sessions during a 12-month period. Parents will also participate in monthly telephone support calls with a Parent Leader during the 12-month intervention period.
  Arms: Intervention

SUMMARY:
The purpose of this study is to 1) convene African American and Latino Community Coalitions to adapt Family Teamwork (FT) for school-age youth, and integrate FT with the Smart and Secure Children (SSC) program community-based, peer delivery format, 2) identify facilitators and barriers to parental involvement in diabetes management for African American and Latino parents of children (5-9 years) with T1D to refine, with Community Coalitions the adapted and integrated Family Teamwork- Peer Delivery (FT-P), and 3) evaluate the feasibility, satisfaction, and preliminary outcomes of the FT-P program among African American and Latino parents of school-aged children (5-9 years) withT1D.

A randomized pilot trials will be conducted with African American and Latino families to examine the feasibility, parent satisfaction, and preliminary outcomes of FT-P. Families will be stratified by race/ethnicity, age, and HbA1c strata, and randomized to FT-P plus standard diabetes care or to standard diabetes care alone after completion of baseline assessment using a random numbers table generated by a program created through Baylor College of Medicine's Institute for Clinical Training and Research data management specialists.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregiver of a child ages 5-10 years with type 1 diabetes as defined by the American Diabetes Association criteria
* Having a child with diabetes duration of >1 year
* Self-identified African American or Latino race/ethnicity
* Fluent in English
* Not planning to leave the geographic area during the study

Exclusion Criterion:

• Not fluent in English

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-05-04 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Intervention Acceptability: Treatment Evaluation Inventory | Immediately post-intervention
  Treatment Evaluation Inventory
Study Enrollment Rate | Pre-Randomization
  Enrollment rate calculated from data obtained from recruitment logs
Study Attrition Rate | 12 months
  Study attrition will be calculated from study logs
Monthly Intervention Calls Completed by Parent Leaders | 12 months
  Percentage of monthly intervention calls completed by Parent Leaders will be determined from study logs

SECONDARY OUTCOMES:
Change in Rate of Average Blood Glucose | Change from baseline at 12 months
  Hemoglobin A1C from medical record
Change in Frequency of Adherence | Change from baseline at 12 months
  Frequency of blood glucose monitoring obtained from blood glucose meter and the Diabetes Self-Management Questionnaire
Change in Level of Child Diabetes Quality of Life: Pediatric Quality of Life Diabetes Module | Change from baseline at 12 months
  Pediatric Quality of Life Total Cumulative Scale (scores range from 0-132 with higher scores indicating worse quality of life)
Change in Level of Parent involvement in diabetes management tasks | Change from baseline at 12 months
  The Diabetes Family Responsibility Questionnaire (scores range from 17-51 with lower scores indicating parent in primarily responsible for diabetes management)
Change in Level of Parent self-efficacy | Change from baseline at 12 months
  Parental Self-Efficacy for Diabetes Management questionnaire scores range from 8-40 with higher scores indicating higher self-efficacy)
Change in Level of Parent diabetes emotional burden | Change from baseline at 12 months
  Problem Areas in Diabetes Revised for Parents (scores range from 0-72 with higher scores indicating less emotional burden)
Change in Level of Parent Depressive Symptoms | Change from baseline at 12 months
  The Center for Epidemiological Depression Studies-Depression scale (scores range from 12-48 with higher scores indicating more depressive symptoms)
Change in Level of Parent Social Support | Change from baseline at 12 months
  2-way Social Support Scale total score (scores range from 0-100 with higher scores indicating more giving and receiving of social support)
Change in Degree of Impact of diabetes on the family system | Change from baseline at 12 months
  Diabetes Family Impact Scale (scores range from 0-56 with higher scores indicating greater impact of diabetes on the family)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley M Butler, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Butler AM, Hilliard ME, Christopher K, Baudino M, Minard C, Karaviti L. Feasibility and acceptability of the TEAM pilot trial with African American and Latino families. J Pediatr Psychol. 2025 May 1;50(5):388-398. doi: 10.1093/jpepsy/jsaf001. PMID 40139919
- See also: PI lab page — https://www.bcm.edu/departments/pediatrics/sections-divisions-centers/psychology/research/health-disparities-laboratory